CLINICAL TRIAL: NCT05841472
Title: An Open-label, Multi-center, Clinical Study to Evaluate Anti-PD-1 Antibody Therapies of Camrelizumab in Combination With Pemetrexed and Carboplatin as First-line Treatment in Patients With Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Anti-PD-1 Antibody Therapies of Camrelizumab in Combination With Pemetrexed and Carboplatin as First-line Treatment in Patients With Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG-SHR-1210-2-01
Record Dates: First submitted 2023-03-30; First posted 2023-05-03 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Non Squamous Non Small Cell Lung Cancer
MeSH Terms: interventions — camrelizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab, Pemetrexed and Carboplatin (Experimental)
  Interventions: Drug: Camrelizumab (SHR-1210), Pemetrexed, and Carboplatin

INTERVENTIONS:
Drug: Camrelizumab (SHR-1210), Pemetrexed, and Carboplatin — * 200 mg of Camrelizumab (SHR-1210) is administered intravenously over a period of around 20-60 min on Day 1 of each 3-week cycle.
  * Pemetrexed 500 mg/m2 is administered intravenously on Day 1 of each 3-week cycle, over a period of more than 10 minutes
  * Carboplatin of AUC 5 is administered intravenously on Day 1 of each 3-week cycle (hydrated as appropriate), over a period of more than 30 minutes by 4-6 cycles.

SUMMARY:
The objective of this bridging study is to acquire new drug approval in Korea for camrelizumab (SHR-1210), a drug that has already been approved in China for treatment in patients with histologically or cytologically confirmed advanced or metastatic (Stage IIIB-IV), EGFR/ALK wild-type, non-squamous, non-small cell lung cancer. In this study, subjects with advanced or metastatic, EGFR/ALK wild-type, non-squamous, non-small lung cancer will receive anti-PD-1 antibody therapy of camrelizumab in combination with pemetrexed + carboplatin as first-line treatment for at least 8 cycles (24 weeks). Then, the best overall RECIST responses (BOR) from subjects who have had at least 1 post-baseline tumor assessment will be evaluated to confirm that camrelizumab, a drug that has already been approved China, has similar efficacy in the Korean population as in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged between 19-80 at the time of signing the informed consent form, male or female.
2. Histologically or cytologically confirmed non-squamous non-small cell lung cancer (NSCLC), Stage IIIB-IV (as per the International Association for the Study of Lung Cancer (IASLC) Staging Handbook in Thoracic Oncology, 8th Edition).
3. The site must provide documented information on EGFR mutation and ALK translocation and both must be negative. Subject cannot be randomized before receiving the source document for EGFR mutation and ALK translocation.
4. A tumor tissue specimen collected upon or after diagnosis of advanced or metastatic disease, either fresh or archival (within 6 months prior to the first dose), must be provided. At least 10 unstained slides can be generated from the formalin fixed, paraffin-embedded (FFPE) tumor tissue block for immunohistochemistry assay or biomarker testing (or may be less than 10 slides as approved by the sponsor's medical monitor). Specimen obtained from fine needle aspiration, pleural fluid smear, or drill biopsy are unacceptable. For bone lesions, specimen without soft tissue components or decalcified bone tumor specimen is also unacceptable.
5. Subjects who have not previously received systemic chemotherapy for advanced/metastatic NSCLC. Chemotherapy as neo-adjuvant/adjuvant therapy or chemoradiotherapy is permitted, as long as the treatment has been completed at least 12 months before the diagnosis of advanced or metastatic disease.
6. Radiographically measurable lesions via CT or MRI, as per RECIST 1.1. The tumor assessment of baseline should be performed within 28 days prior to the first dose.
7. ECOG PS score: 0-1.
8. Expected survival ≥ 3 months.
9. Subjects must undergo all screening laboratory tests as per the protocol within 14 days prior to the first dose. Laboratory tests at screening must meet the following criteria:

1) Hematology: (without blood transfusion, G-CSF, or medication within 14 days prior to screening)

1. Hemoglobin (HB) ≥ 90 g/L;
2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L;
3. Platelet (PLT) ≥ 100 x 109/L;
4. White blood cell (WBC) ≥ 4.0 x 109/L and ≤ 15 x 109/L; 2) Biochemistry: (no blood or albumin transfusion within 14 days prior to screening)
5. AST and ALT ≤ 1.5 x ULN (≤ 5 x ULN for liver metastasis);
6. ALP ≤ 2.5 x ULN (≤ 5 x ULN for bone metastasis);
7. TBIL ≤ 1.5 x ULN;
8. ALB ≥ 30 g/L;
9. Cr ≤ 1.5 x ULN, and creatinine clearance (CrCL) ≥ 60 mL/min (Cockcroft-Gault equation);
10. APTT ≤ 1.5 x ULN, and INR or PT ≤ 1.5 x ULN (no anticoagulant therapy).

    10. Female subjects of childbearing potential must have a negative serum pregnancy test within 3 days prior to the first dose. Female subjects of childbearing potential and male subjects with partners of childbearing potential must agree to use adequate method of contraception during the study period and 180 days after the last dose of study medication.

    11. Subject has voluntarily agreed to participate by giving written informed consent/assent.

    Exclusion Criteria:

    1. Exclusion criteria for the target indication
    1. Subjects with other histological types besides non-squamous non-small cell lung cancer, including mixed carcinomas or NSCLC with small cell lung cancer components/neuroendocrine differentiation.
    2. Subjects with EGFR mutation or ALK translocation.
    3. Subjects without radiographically measurable lesions.
    4. Subjects with carcinomatous meningitis and spinal cord compression.
    5. Subjects with untreated central nervous system (CNS) metastasis. Subjects with previously treated CNS metastases may participate if the CNS metastasis is limited to the supraentorial and cerebellar regions, adequately treated, and clinically stable (by radiological tumor assessments, preferably enhanced MRI or CT) for at least 4 weeks, and if the subject's neurological symptoms can return to NCI-CTCAE Grade ≤ 1 within 2 weeks prior to the first dose. In addition, subjects who are using corticosteroids for clinical symptoms are not eligible, unless the doses of corticosteroids stable or gradually reduced to prednisone ≤ 10 mg/day (or equivalent) -for at least 2 weeks.
    6. Subjects who can be treated with surgical resection or radical radiotherapy.
    7. Subjects who previously received treatment with any other anti-PD-1(L1) or CTLA4 monoclonal antibodies.

    2. Medical history and complications
    1. Subjects with any active, known, or suspected autoimmune diseases. Subjects who are clinically stable and do not require systemic immunosuppressants, such as those with Type I diabetes, hypothyroidism requiring only hormone replacement therapy, or skin diseases that do not require systemic treatment (for example, vitiligo, psoriasis or alopecia), or subjects in whom recurrence are not expected without external triggers may be eligible.
    2. Subjects with any complication that require systemic corticosteroids like prednisone (> 10 mg/day or equivalent) or other immunosuppressants within 14 days prior to the first dose. In the absence of active autoimmune disease, inhaled or topical use of corticosteroids, and physiologic hormone replacement therapy for adrenal insufficiencylike prednisone > 10 mg/day or equivalent are permitted;
    3. Subjects who received cancer vaccines or other immunostimulatory anti-cancer agents (interferon, interleukin, thymosin, or immune cell therapy) within 1 month prior to the first dose.
    4. Subjects who are currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks (or 5 half-lives of the previous investigational agent) prior to the first dose.
    5. Subjects who are expected to require any other forms of anti-cancer treatment (including maintenance treatment with other drugs, radiotherapy, and/or surgical resection) for NSCLC while on study.
    6. Subjects who received major surgery within 4 weeks prior to the first dose, non-thoracic radiation therapy > 30 Gy within 4 weeks prior to the first dose, thoracic radiation therapy > 30 Gy within 24 weeks prior to the first dose, or palliative radiation ≤ 30 Gy within 2 weeks prior to the first dose, and failed to recover from the toxicities and/or complications of these interventions to NCI-CTC AE Grade ≤ 1 (except for alopecia and fatigue). Palliative radiotherapy for symptomatic control is permitted, but must be completed within 2 weeks prior to the first dose and no additional radiotherapy should be scheduled for the same lesion.
    7. Subjects highly suspected of interstitial lung disease, or with conditions that may interfere with the testing or management of suspected treatment-related pulmonary toxicities, or other moderate to severe lung diseases that seriously affect pulmonary function.
    8. Subjects who require concomitant treatment for other active malignant tumors.
    9. Subjects with a history of prior malignant tumors, except for basal cell carcinoma, superficial bladder cancer, squamous cell carcinoma of the skin, or cervical carcinoma in situ with complete remission for at least 5 years prior to screening and no additional treatment is required or expected while on study.
    10. Subjects with Grade II or higher myocardial ischemia or myocardial infarction, or poorly controlled arrhythmias. Subjects with NYHA Class III-IV cardiac insufficiency or an LVEF (left ventricular ejection fraction) < 50% by echocardiography.
    11. Subjects with significant hemoptysis or coughing a daily volume up to half a teaspoon (2.5 mL) or more of blood within 1 month prior to randomization.
    12. Subjects with clinically significant hemorrhage or clear bleeding tendency within 1 month prior to randomization, such as GI bleeding, hemorrhagic gastric ulcer, or vasculitis.
    13. Events of arterial/venous thrombosis within 3 months prior to randomization, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, brain infarction), deep vein thrombosis, and pulmonary embolism.
    14. Subjects with active pulmonary tuberculosis (TB). Active TB should be ruled out in subjects suspected of such condition, by chest X-ray, sputum test, and examinations of clinical symptoms and signs. Subjects with a history of active TB infection within 1 year prior to the screening are excluded, despite being treated. Subjects with a history of active TB infection more than 1 year ago can be enrolled if the course and type of TB treatment are appropriate.
    15. Subjects with serious infection within 4 weeks prior to the first dose, including but not limited to infective complications, bacteremia and severe pneumonia that require hospitalization. Subjects with any active infections are excluded, lymphangitic spread of the NSCLC is not exclusionary.
    16. Subjects who prepare to receive or have previously received tissue/organ transplants.
    17. Subjects who plan to receive or have received live vaccines within 30 days prior to the first dose.
    18. Subjects with contraindications for platinum-based medications before the first dose: gout, varicella, herpes zoster, and Grade ≥ 2 peripheral neuropathy.
    19. It is not recommended to enroll subjects with uncontrolled tumor-related pain. Subjects requiring pain medication must have a stable regimen before randomization. Palliative radiotherapy for symptomatic lesions (such as bone metastasis or perineural invasion) should be completed at least 2 weeks before enrollment. Loco-regional treatment should be considered before randomization, if appropriate, for asymptomatic metastatic lesions where further growth may result in functional deficits or intractable pain (e.g., epidural metastasis without spinal cord compression).

    3. Physical examination and laboratory tests
    1. Subjects have known history of human immunodeficiency virus (HIV) seropositive status or acquired immunodeficiency syndrome (AIDS).
    2. Subjects with untreated active hepatitis. Hepatitis B: Hepatitis B surface antigen (HBV sAg) positive and HBV DNA greater than the upper limit of normal; Hepatitis C: HCV antibody (HCV Ab) positive and HCV RNA positive, and abnormal hepatic function; Hepatitis B and C coinfection.
    3. Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.

    4. Allergies and adverse drug reactions
    1. Severe allergic, anaphylactic, or other hypersensitivity reactions to other monoclonal antibodies.
    2. Allergy or intolerance during an infusion.
    3. History of severe allergies to pemetrexed, carboplatin, or their premedications.

    5. Subjects with mental illness, alcohol abuse, inability to quit smoking, and drug or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

    6. Based on the investigator's opinion, subjects with a history or current evidence of any condition, diseases, treatments, or laboratory abnormalities that may confound the study results, interfere with study procedures, or are not in the best interests of the subjects, should be excluded.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Best overall RECIST response, BoR | up to 8 cycles (24 weeks) of the last subject

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 6 months, 12 months, 24 months
Objective response rate (ORR) | 6 months, 12 months, 24 months
Overall survival (OS) | up to 6 months from the last visit of the last patient
Disease control rate (DCR) | 6 months, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Lee, MD, Principal Investigator — Korea University Guro Hospital
Locations (8):
- South Korea (8):
  - Korea University Anam Hospital, Anam
  - Hallym University Sacred Heart Hospital, Anyang
  - Chonnam National University Hwasun Hospital, Hwasun
  - Catholic University of Korea EunPyeong St. Mary's Hospital, Seoul
  - Catholic University of Korea Yeouido St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul Asan Hospital, Seoul
  - Busan National University Hospital Yangsan, Yangsan